CLINICAL TRIAL: NCT05199792
Title: Efficacy of Gadoterate Meglumine in Diagnosis of Vascular Diseases Using MRA
Brief Title: Efficacy of Gadoterate Meglumine in Diagnosis of Vascular Diseases Using MRA MRA
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, James Carr, Professor, Northwestern University
Other Study IDs: STU00205041
Record Dates: First submitted 2021-12-08; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2x dose of Dotarem: qualifying MRA
  Interventions: Diagnostic Test: Dotarem

INTERVENTIONS:
Diagnostic Test: Dotarem — (Dotarem) (0.4 ml/kg (0.2 mmol/kg))

SUMMARY:
The purpose of this study is to compare magnetic resonance angiography (MRA) using gadoterate meglumine to clinically obtained MRA using gadobutrol. The specific aims are to show:

1. Carotid, chest, and abdomenal MRA with gadoterate meglumine has a comparable image quality and diagnostic confidence to MRA using gadobutrol.
2. Carotid, chest, and abdomenal MRA with gadoterate meglumine has a comparable accuracy for vascular lesion and stenosis detection compared to MRA using gadobutrol.

DETAILED DESCRIPTION:
In this study, we will assess the image quality and accuracy of MRA studies acquired using these two contrast agents. In the cases where Digital Subtraction Angiography (DSA) or CT angiography images are available, the results of the study using both contrast agents will be compared to the DSA or CTA findings. All MRA images will be assessed independently by two readers. The readers will be blinded to the clinical symptoms, contrast agent and DSA/CTA results. A five-level system rating for image quality of each arterial segment will be used (1 = non-diagnostic images, 2 = poor image quality, significant blurring/artefacts, diagnosis suspected but not established, 3 = fair quality with established diagnosis, 4=good quality with definite diagnosis, minimal blurring/artefacts, 5 = sharply defined borders, excellent quality image information). Vascular lesions will also be graded on a 1-5 scale. Vessel segment stenoses will be graded using a five-point grading scale as follows: (1) normal; (2) mild (<50% diameter stenosis); (3) moderate (50% to 74%), severe (75% to 99%); and (5) total occlusion.

Grades 1 and 2 will be considered insignificant, while grades 3 to 5 will be interpreted as significant for diagnostic accuracy testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-89 years of age
* Suspected or diagnosed vascular disease
* Standard of care carotid, chest, or
* Willingness to undergo 1 research MRA with up to double dose gadoterate meglumine
* Able to complete the MR safety questionnaire
* Able to comprehend and provide informed consent in English

Exclusion Criteria:

* • Allergy to gadolinium-containing contrast media

  * Chronic, severe kidney disease
  * eGFR < 60mL/min/1.73m2
  * Acute kidney injury
  * Kidney or liver transplant within 8 weeks
  * Contraindication to MRI (implanted device, claustrophobia, dyspnea precluding the ability to follow breath-hold instructions)
  * Pregnant or breastfeeding women
  * Adults unable to consent
  * Individual who are not yet adults
  * Prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: qualifying MRA
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of MRA image quality | 18 months
  assess the image quality of MRA studies acquired using these two contrast

SECONDARY OUTCOMES:
Assessment of MRA accuracy | 18 months
  Assess the accuracy of MRA studies acquired using these two contrast

CONTACTS AND LOCATIONS:
Overall Officials: James Carr, Principal Investigator — Northwestern University
Locations (1):
- Yasmeen Khan, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eng J. Sample size estimation: how many individuals should be studied? Radiology. 2003 May;227(2):309-13. doi: 10.1148/radiol.2272012051. PMID 12732691
- [Result] Seeger A, Kramer U, Fenchel M, Grimm F, Bretschneider C, Doring J, Klumpp B, Tepe G, Rittig K, Seidensticker PR, Claussen CD, Miller S. Comparison between a linear versus a macrocyclic contrast agent for whole body MR angiography in a clinical routine setting. J Cardiovasc Magn Reson. 2008 Dec 30;10(1):63. doi: 10.1186/1532-429X-10-63. PMID 19116027